CLINICAL TRIAL: NCT00458926
Title: Enhancing Utilization of Non-Invasive Positive Pressure Ventilation in Critical Care
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 6742
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: COPD; Congestive Heart Failure; Asthma; Respiratory Distress Syndrome, Adult; Pneumonia
Keywords: ventilation, mechanical; intubation, endotracheal; respiratory insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Asthma; Respiratory Distress Syndrome; Pneumonia; Respiratory Aspiration; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-invasive positive pressure ventilation (NIV) refers to the provision of mechanical ventilation without an artificial airway (for example, an endotracheal tube). Over the past decade, evidence from randomized control trials has accumulated to demonstrate effectiveness of the technique in avoiding intubation, reducing complications associated with intubation, shortening ICU and hospital lengths of stay, and reducing mortality rates in selected patients with acute respiratory failure. However, NIV is still underutilized at many medical centers. The purposes of this project will be to acquire information related to NIV use, to identify reasons for underutilization, to implement interventions that encourage more appropriate use of NIV, and to evaluate the effectiveness of the interventions. Reliable information on NIV use as well as analysis of reasons for underutilization will provide insight into ways of enhancing NIV use. We will determine utilization rate, technology used, patient diagnoses, duration of ventilator use and hospital stay, and success rates as recorded on case report forms (CRFs). After completing the survey, we will provide an educational program to randomly selected institutions (one-half of the total) aimed at increasing the knowledge and skill of physicians, nurses, and therapists regarding use and implementation of NIV. Data will be gathered for a second round with the same data-gathering instruments used during

DETAILED DESCRIPTION:
Project Focus The focus of this project is to improve the ventilatory management of patients with acute respiratory failure in the critical care setting by enhancing the use of non-invasive ventilation, a goal that should lead to improved outcomes and efficiency of care. Within the framework of the funding agency, the Chest Foundation, this proposal aims to promote the use of alternative therapies in treating patients with critical illness, educate practitioners, and disseminate new knowledge regarding the therapy.

Background Non-invasive positive pressure ventilation (NPPV) provides mechanical ventilation without the need for airway invasion through the use of either nasal or oronasal masks (covering both the nose and mouth) attached to positive pressure ventilators. Published evidence from randomized control trials has demonstrated the effectiveness of the technique in avoiding intubation, reducing complications associated with intubation, shortening ICU and hospital lengths of stay, and reducing mortality rates in selected patients with acute respiratory failure. Randomized trials have demonstrated effectiveness in patients with acute exacerbations of COPD (1-3), cardiogenic pulmonary edema (4), immunocompromised patients with hypoxemic respiratory failure (5,6), facilitating the weaning process in patients ventilated invasively (7), and in patients who develop respiratory insufficiency after lung resection (8). In addition, evidence that is not quite as strong supports the use of NPPV in patients with acute asthma (9), cystic fibrosis (10), community-acquired pneumonia if there is underlying COPD (11), and patients with a do-not-intubate status (12).

Based on this evidence, consensus groups have recommended the use of NPPV in treating patients with COPD exacerbations and for selected patients with other diagnoses (13). However, NPPV is still underutilized at many medical centers throughout the world (14) and it is fair to presume that many patients are being deprived of NPPV's advantages and that ICU resources are being wasted. Similar surveys have not been performed in the US, and my firm impression from polling audiences when I speak on this subject is that a similar proportion of US centers are not using NPPV. The purposes of this project are to acquire this information in a US setting, to identify reasons for underutilization, to implement interventions that encourage more appropriate use of NPPV, and then to evaluate the effectiveness of the intervention.

The successful implementation of this project may have a major impact on the practice of critical care medicine. Reliable information on utilization of NPPV as well as analysis of reasons for underutilization will provide insight into ways of enhancing utilization. Educational programs designed to enhance practitioners' skills in implementing NPPV should lead to greater utilization and improved success rates. Optimal utilization of NPPV should lead to improved outcomes for patients with respiratory failure, more rational use of resources, and lower ICU costs for our health care system.

Project A. Major Hypothesis: An educational intervention will increase utilization and success rates of NPPV in hospitals that currently underutilizing it.

B. General Outline 1. Site selection

1. Select 8 sites that use NPPV in < 10% of patients receiving mechanical ventilatory assistance, based on a survey mailed to acute care hospitals in Massachusetts and Rhode Island during 2002. Sites will be selected based on: (i) willingness to participate (as per request of Respiratory Therapy director), (ii) > 30 mechanical ventilation initiations/month as reported in the survey, and (iii) n more than 90 minute drive from Boston.
2. Perform prospective evaluation of use of NPPV that will determine rate of utilization, technology used, patient diagnoses, duration of ventilator use and hospital stay, and success rates as recorded on case report forms.
3. Intervention (or control) phase. After completion of survey, provide education/in-servicing program to 5 randomly selected sites aimed at increasing knowledge and skill of physicians, nurses, and respiratory therapists in the use and implementation of NPPV.

   C. Evaluation phase

   1. Re-survey targeted institutions with regard to use of NPPV and patient outcomes.

   Methods A. Prospective Survey at 8 Selected Institutions Underutilize NPPV
   1. Random selection will be performed using computer-generated number sequence, selecting sites based on alphabetical listing.
   2. Data will be gathered on CRFs that will document utilization of mechanical ventilation; number of NPPV starts; patient diagnoses; date, time, and location of NPPV use; equipment and settings used to ventilate; success rate of NPPV; duration of NPPV use; and eventual patient outcomes.
   3. Data collectors from Tufts or respiratory therapists at each site will initiate CRF use. Personal health information will be de-identified by using study code numbers. The patient medical record number cross-referenced to the patient code will be kept on a separate list kept in a locked area, so that the patient's medical record can be located to retrieve missing data and recorded data can be verified.

   B. Education and In-Servicing

   Educational and in-servicing sessions will be provided to randomly selected underutilizing sites and will review guidelines provided in the literature by the PI (15,16) as well as other investigators (17). Grand rounds and other lecture venues for the physicians working in emergency and critical care settings will describe the skills needed to select patients who will benefit from the use of NPPV. Workshops for respiratory therapists will review patient selection, proper use of equipment, and monitoring and weaning techniques. In-servicing sessions for emergency and critical care nurses will review the rationale behind NPPV use and how to monitor patients who are placed on NPPV. At control sites, no intervention will be undertaken prior to the second data survey.

   C. Evaluation Phase

   Mechanical ventilation and NPPV utilization will be tracked with the same data gathering instruments used during the initial phase. Initial and follow-up data gathering will be staggered. The follow-up evaluation in the control group will be timed to correspond with follow-up in institutions receiving the intervention.

   Main Outcome Variables
   1. Rate of NPPV utilization.
   2. NPPV success.
   3. Compliance with guidelines.

   Analysis The main outcome variables will be analyzed as categorical variables by chi square analysis or the Mann-Whitney test as appropriate. Initial data will be compared to follow-up data obtained during the follow-up phase using paired t-tests, Mann-Whitney tests, as appropriate. Comparisons between the intervention and control groups at baseline and follow-up will be made using unpaired t-tests or chi square analyses as appropriate. Because randomization is by site, data will be clustered by institution, although we will be limited by resources as to the number of sites in this study. Using linear regression analysis, we will be able to determine risk ratios for failure for a number of initial characteristics, including diagnosis, vital signs, blood gases, presence of cough and airway secretions, body mass index, sedation, kind of equipment used, in-hospital locations for NPPV implementation, and other characteristics.

   Anticipated Results We anticipate that results from the sites selected to receive the training intervention and control sites will be similar at baseline and that the intervention will increase utilization and success rates of NPPV compared to baseline. Utilization and training rates also may increase at control sites, because of an increased trend toward NPPV use in acute care settings. However, the important comparison will be between the intervention and control sites at follow-up. If intervention is effective, NPPV utilization and success rates will be increased at intervention sites compared to controls. Other key differences may be detectable, such as shorter ICU lengths of stay and reduced mortality rates among respiratory failure patients treated at the intervention sites.

   Risk/Benefit Analysis This is a prospective observational trial that involves no patient intervention. Patients are to be managed by their primary caregivers, and guidelines are provided to randomly selected institutions. These guidelines, derived from standards in the literature (15-17) aim to improve the outcomes of patients receiving NPPV. Because the trial is observational, involves no direct patient intervention, and poses essentially no direct risk to patients, we are requesting waiver of consent. The patient data that we are collecting aims to track standard clinical information and will be de-identified.

   Protection of Personal Health Information CRFs will be de-identified for the purposes of the study. CRFs will be kept in a locked office. A cross-referenced sheet containing medical record numbers and patient code numbers will be kept in a locked file until missing data are retrieved and data verified using chart review. Once the data set is complete and validated, the cross-referenced sheet will be shredded and discarded.

   Limitations, Potential Problems, and Strengths One limitation is that optimal utilization rates for NPPV in the acute care setting have not been established. In addition, overutilization (use in inappropriate candidates) at some centers is also a concern, as noted in the European survey (14). Although this project will focus on underutilization of NPPV, we will able to track evidence of inappropriate applications. Another concern is that there can be no blinding as to study condition at individual centers, introducing the possibility of center-based bias. Randomization of intervention and control centers should minimize this concern.

   The study also has several strengths. Compared to the European ICU survey that only included selected centers that had volunteered to serve in a consortium, this project will obtain information on NPPV use in all acute care centers in a geographic region, giving a more accurate glimpse of actual usage rates. In addition, the survey will provide information on reasons for under-utilization and the inclusion of an intervention will shed light on the effectiveness of strategies to enhance utilization. These results can then be applied to achieve more appropriate use of NPPV. The study might also provide insight into techniques that could also be applied to other critical care practices, such as use of particular ventilator settings for invasive mechanical ventilation, or use of certain pharmacological agents.

   References
   1. Kramer N, Meyer TJ, Meharg J et al: Randomized, prospective trial of noninvasive positive pressure ventilation in acute respiratory failure. Am J Respir Crit Care Med 1995; 151: 1799-1806.
   2. Brochard L, Mancebo J, Wysocki M et al: Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med 1995; 333: 817-822.
   3. Plant PK, Owen JL, and Elliott MW: Early use of noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease on general respiratory wards: a multicenter randomized controlled trial. Lancet 2000; 355:1931-1935.
   4. Masip J, Betbese AJ, Paez J, Vecilla F, Canizares R, Padro J, Paz Marco A, Otero J, Bllus J: Non-invasive pressure support ventilation versus conventional oxygen therapy in acute cardiogenic pulmonary oedema; a randomized study. Lancet 2000; 356:2126-2132.
   5. Antonelli M, Conti G, Bufi M, Costa MG, Lappa A, Rocco M, Gasparetto M, Meduri GU: Noninvasive ventilation for treatment of acute respiratory failure in patients undergoing solid organ transplantation. JAMA 2000, 283: 235-241.
   6. Hilbert G, Gruson D, Vargas F, Valentino R, Gbikpi-Benissan G, Dupon M, Reiffers J, and Cardinaud JP. Noninvasive ventilation in Immunosuppressed patients with pulmonary infiltrates, and acute respiratory failure. N Engl J Med 2001; 344:481-487.
   7. Nava S, Ambrosino N, Clini E, Prato M, Orlando G, et al. Non-invasive mechanical ventilation in the weaning of patients with respiratory failure due to chronic obstructive pulmonary disease: a randomized study. Ann Intern Med 1998; 128: 721-728.
   8. Auriant I, Jallot A, Herve P, et al. Noninvasive ventilation reduces mortality in acute respiratory failure following lung resection. Am J Respir Crit Care Med 2001; 164: 1231-1235.
   9. Meduri GU, Cook TR, Turner RE, Cohen M and Leeper KV. Noninvasive positive pressure ventilation in status asthmaticus. Chest 1996; 110: 767-774
   10. Hodson ME, Madden BP, Steven MH et al. Noninvasive mechanical ventilation for cystic fibrosis patients - a potential bridge to transplantation. Eur Respir J 1991; 4: 524-527.
   11. Confalonieri M, Potena A, Carbone G, Della Porta R, Tolley EA, and Meduri GU. Acute respiratory failure in patients with severe community-acquired pneumonia. Am J Respir Crit Care Med 1999, 160: 1585-1591.
   12. Meduri GU, Fox RC, Abou-Shala N, et al. Noninvasive mechanical ventilation via face mask in patients with acute respiratory failure who refused endotracheal intubation. Crit Care Med 1994; 22: 1584-1590.
   13. Bach JR, Brougher P, Hess DR et al. Consensus statement: Noninvasive positive pressure ventilation. Respir Care 1997; 42: 365-369. 6. 6.
   14. Carlucci A, Richard J-C, Wysocki M, Lepage E, Brochard L. Noninvasive versus conventional mechanical ventilation: and epidemiological survey. Am J Respir Crit Care Med 2001; 163:874-880.
   15. Criner GJ, Kreimer DT, Tomaselli M, Pierson W, and Evans D. Financial implications of noninvasive positive pressure ventilation (NPPV). Chest 1995; 108: 475-481.
   16. Hill NS, ed. Noninvasive Positive Pressure Ventilation; Principles and Applications. Futura, Armonk, NY, 2001.
   17. Sinuff T, Cook DJ, Randall J, Allen CJ. Evaluation of a practice guideline for noninvasive positive pressure ventilation for acute respiratory failure. Chest 2003; 123(6):2062-73.

ELIGIBILITY:
Inclusion Criteria:

* Starting on mechanical ventilation (including: invasive, noninvasive, CPAP or BiPAP for purpose of treatment of respiratory failure)
* 18 years of age or older

Exclusion Criteria:

* Use of home mechanical ventilation, including nocturnal ventilation, continuous mechanical ventilation,BiPAP.
* Continuous use of CPAP or BiPAP for treatment of obstructive sleep apnea.
* Placed on mechanical ventilation for purposes of surgical anesthesia or use of anesthesia for a diagnostic procedure.
* Patient has tracheostomy or was intubated endotracheally prior to admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who require mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2003-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S. Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ozsancak Ugurlu A, Sidhom SS, Khodabandeh A, Ieong M, Mohr C, Lin DY, Buchwald I, Bahhady I, Wengryn J, Maheshwari V, Hill NS. Use and Outcomes of Noninvasive Ventilation for Acute Respiratory Failure in Different Age Groups. Respir Care. 2016 Jan;61(1):36-43. doi: 10.4187/respcare.03966. Epub 2015 Sep 15. PMID 26374908
- [Derived] Ozsancak Ugurlu A, Sidhom SS, Khodabandeh A, Ieong M, Mohr C, Lin DY, Buchwald I, Bahhady I, Wengryn J, Maheshwari V, Hill NS. Where is Noninvasive Ventilation Actually Delivered for Acute Respiratory Failure? Lung. 2015 Oct;193(5):779-88. doi: 10.1007/s00408-015-9766-y. Epub 2015 Jul 26. PMID 26210474
- [Derived] Ozsancak Ugurlu A, Sidhom SS, Khodabandeh A, Ieong M, Mohr C, Lin DY, Buchwald I, Bahhady I, Wengryn J, Maheshwari V, Hill NS. Use and outcomes of noninvasive positive pressure ventilation in acute care hospitals in Massachusetts. Chest. 2014 May;145(5):964-971. doi: 10.1378/chest.13-1707. PMID 24480997